CLINICAL TRIAL: NCT00111059
Title: Cross-Sectional Case-Control Study on Obesity, Cardiovascular and Psycho-Social Characteristics in the City of Merzig
Brief Title: Primary Prevention Study: Study on Obesity, Cardiovascular and Psycho-Social Characteristics in the City of Merzig
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Other Study IDs: 1
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Obesity; Cardiovascular Disease; Depression; Stress
Keywords: obesity; cardiovascular disease; depression; stress
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Cardiovascular risk factors and psycho-social characteristics will be determined in obese and non-obese patients in the setting of primary medical care.

DETAILED DESCRIPTION:
Cardiovascular risk factors and psycho-social characteristics will be determined using a questionnaire in primary care physician offices in the city of Merzig, Germany. We will recruit all people (age>18y) with a body-mass index (BMI) > 30 kg/m2 plus patients in the two following participating physician offices: Praxisnetz and Merzig. Cardiovascular risk will be assessed using the PROCAM (Munster Heart Study), ESC (European Society of Cardiology) and Framingham risk scores. Psycho-social factors will be recorded according to the methodology of the INTERHEART study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or > 18
* BMI > 30 kg/m2
* Presenting to a participating primary care physician

Exclusion Criteria:

* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-01; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Klinik Innere Medizin III, Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Praxisnetz Merzig, Merzig, Saarland

REFERENCES:
- [Background] Assmann G, Cullen P, Schulte H. Simple scoring scheme for calculating the risk of acute coronary events based on the 10-year follow-up of the prospective cardiovascular Munster (PROCAM) study. Circulation. 2002 Jan 22;105(3):310-5. doi: 10.1161/hc0302.102575. PMID 11804985
- [Background] Rosengren A, Hawken S, Ounpuu S, Sliwa K, Zubaid M, Almahmeed WA, Blackett KN, Sitthi-amorn C, Sato H, Yusuf S; INTERHEART investigators. Association of psychosocial risk factors with risk of acute myocardial infarction in 11119 cases and 13648 controls from 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):953-62. doi: 10.1016/S0140-6736(04)17019-0. PMID 15364186